CLINICAL TRIAL: NCT00824473
Title: Randomized, Double-Blind, Placebo-Controlled Trial of the Safety and Efficacy of MP03-36 in Subjects With Seasonal Allergic Rhinitis
Brief Title: A Study to Evaluate the Safety and Effectiveness of a Nasal Spray to Treat Seasonal Allergies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Meda Pharmaceuticals (Industry)
Responsible Party: Harry Sacks, MD Vice President, Medical and Scientific Affairs, Meda Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MP443
Record Dates: First submitted 2009-01-14; First posted 2009-01-16 (Estimated); Results first posted 2010-01-28 (Estimated); Last update posted 2010-02-23 (Estimated); Status verified 2010-02

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — azelastine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- 2 (Active Comparator): 0.15% azelastine hydrochloride
  Interventions: Drug: 0.15% azelastine hydrochloride

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: 1
Drug: 0.15% azelastine hydrochloride — 0.15% azelastine hydrochloride 822 mcg
  Arms: 2

SUMMARY:
The purpose of this study is to determine if one allergy medication (0.15% azelastine hydrochloride) is more effective than Placebo alone

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects 12 years of age and older
2. Provide written informed consent/pediatric assent. If the subject is a minor, a parent or legal guardian must give written informed consent
3. Screening Visit: Have a 12-hour reflective TNSS of at least 8 out of a possible 12 and a congestion score of 2 or 3 on visit 1
4. Randomization Visit: Have a 12-hour reflective TNSS (AM or PM) of at least 8 on 3 separate symptom assessments (one of which was within 2 days of visit 2, and can include the morning of visit 2) during the Lead-in Period. In addition, an AM or PM 12-hour reflective nasal congestion score of 2 or 3 must have been recorded on 3 separate symptom assessments (one of which was within 2 days of visit 2, and can include the morning of visit 2)
5. Willing and able to comply with the study requirements
6. At least a 2-year history of SAR during Texas Mountain Cedar season
7. The presence of IgE-mediated hypersensitivity to Texas Mountain Cedar, confirmed by a positive response to skin prick within the last year. A positive response is defined as a wheal diameter of at least 3 mm larger than the negative control.
8. General good health and free of any disease or concomitant treatment that could interfere with the interpretation of the study results as determined by the investigator or the sponsor's medical officer. When in doubt, the investigator should confer with the sponsor's medical monitor or designee to determine eligibility for the study.
9. Subjects receiving immunotherapy injections (antigen desensitization) must be on a stable maintenance regimen for at least 30 days before the first study visit (adjustments to regimen following a brief period of missed injections do not preclude participation).Dose reduction when a new bottle is used does not preclude participation.
10. Subjects currently receiving sublingual immunotherapy are excluded. A 6-month washout period is required following the last dose of sublingual immunotherapy.

Exclusion Criteria:

1. On Focused Nasal Examination, the presence of any superficial and moderate nasal mucosal erosion, nasal mucosal ulceration, or nasal septum perforation (Grade 1b-4) at either screening visit or randomization visit will disqualify the subjects from the study.
2. Other nasal disease(s) likely to affect deposition of intranasal medication, such as sinusitis, rhinitis medicamentosa, clinically significant polyposis, or clinically significant nasal structural abnormalities.
3. Nasal surgery or sinus surgery within the previous year.
4. Chronic sinusitis - more than 3 episodes per year
5. Planned travel outside of the study area during the study period
6. The use of any investigational drug within 30 days prior to visit 1. No investigational products are permitted for use during the conduct of this study
7. Presence of any hypersensitivity to drugs similar to azelastine and to either sorbitol or sucralose (Splenda® brand sweetener)
8. Women who are pregnant or nursing
9. Women of childbearing potential who are not abstinent or not practicing a medically acceptable method of contraception
10. Respiratory Tract Infections within 14 days prior to visit 1
11. Respiratory Tract Infections requiring antibiotic treatment 14 days prior to visit 1
12. Asthma (with the exception of intermittent asthma). Subjects with mild, intermittent asthma who only require short-acting inhaled bronchodilators (not more often than twice per week) and who do not have nocturnal awakening as a result of asthma are eligible for enrollment
13. Significant pulmonary disease including COPD
14. Clinically significant arrhythmia or symptomatic cardiac conditions
15. A known history of alcohol or drug abuse within the last 2 years
16. Existence of any surgical or medical condition or physical or laboratory findings, which in the opinion of the investigator or sponsor's medical monitor, might significantly alter the absorption, distribution, metabolism, or excretion of study drug; that might significantly affect the subject's ability to complete this trial; or their safety in this trial.
17. Clinically relevant abnormal physical findings within 1 week of randomization which, in the opinion of the investigator, would interfere with the objectives of the study or that may preclude compliance with the study procedures
18. Participation in MedPointe Protocols MP439 or MP440.
19. Employees of the research center / private practice and their family are excluded

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 506 (Actual)
Dates: Start 2008-12; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lewis M Fredane, MD, Study Director — Meda Pharmaceuticals
Locations (7):
- United States (7):
  - Allergy and Asthma Associates, Austin, Texas
  - Allergy and Asthma Center of Austin, Austin, Texas
  - Central Texas Health Research, New Braunfels, Texas
  - Southwest Allergy and Asthma Center, P.A., San Antonio, Texas
  - Sylvana Research Associates, San Antonio, Texas
  - Allergy, Asthma Research Center, San Antonio, Texas
  - Allergy and Asthma Center, Waco, Texas

REFERENCES:
- [Derived] Howland WC, Amar NJ, Wheeler W, Sacks H. Efficacy and safety of azelastine 0.15% nasal spray administered once daily in patients with allergy to Texas mountain cedar pollen. Int Forum Allergy Rhinol. 2011 Jul-Aug;1(4):275-9. doi: 10.1002/alr.20065. Epub 2011 May 9. PMID 22287431

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First observation: 30 Dec 2008 Last observation: 13 Feb 2009
Pre-assignment Details: Subjects participated in a 7 day screening period to Identify appropriate subjects based on symptom scores.
Groups:
- Placebo: Placebo Nasal Spray/2 sprays per nostril once a day for 14 days
- Astepro 0.15%: 0.15% azelastine hydrochloride Nasal Spray/2 sprays per nostril once a day for 14 days
Period: Overall Study
Arm/Group | Placebo | Astepro 0.15%
Started | 255 (1 subject was randomized in error) | 251
Completed | 240 | 238
Not Completed | 15 | 13
Not completed — Adverse Event | 4 | 5
Not completed — Lack of Efficacy | 2 | 2
Not completed — Protocol Violation | 2 | 0
Not completed — Non-Compliance | 4 | 2
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Other | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Astepro 0.15% | Total
Number analyzed (Participants) | 254 | 251 | 505
Age, Categorical [Count of Participants; unit: Participants] — Number of participants based on ITT population
  Participants
    <=18 years | 27 | 24 | 51
    Between 18 and 65 years | 220 | 218 | 438
    >=65 years | 7 | 9 | 16
Age Continuous [Mean (Standard Deviation); unit: years] — Number of participants based on ITT population
  years | 38.5 (14.59) | 38.0 (14.40) | 38.2 (14.48)
Sex: Female, Male [Count of Participants; unit: Participants] — Number of participants based on ITT population
  Participants
    Female | 150 | 157 | 307
    Male | 104 | 94 | 198
Region of Enrollment [Number; unit: participants] — Number of participants based on ITT population
  participants
    United States | 254 | 251 | 505

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 12-hour Reflective Total Nasal Symptom Score(rTNSS)for the Entire 14-day Study Period Compared to Placebo (AM and PM Combined)at 14 Days
Description: rTNSS consisting of runny nose, itchy nose, nasal congestion, and sneezing was assessed twice daily. Each symptom is rated on a scale from 0-3: 0=none, 1=mild, 2=moderate, and 3=severe. (maximum 12 points per assessment.) Total possible score is 24 per day.
  Least square means was controlled for study day as the within-patient effect, treatment group and site as the between-patient effects, treatment by-study day interaction, and basline as a covariate.
Time Frame: baseline and 14 days
Measure: Least Squares Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Astepro 0.15%
Number analyzed (Participants) | 255 | 251
Scores on a scale
  Baseline symptom score | 18.76 (3.301) | 18.48 (3.231)
  Overall change from baseline | -2.14 (3.696) | -3.57 (4.242)
Statistical Analysis 1: Comparison: Placebo vs Astepro 0.15%; Overall change from baseline; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA is being used due to a covariate being included in the model. The covariate is baseline TNSS score; Mean Difference (Final Values) = -1.4286, 95% CI [-2.12 to -0.74], Standard Error of Mean 0.3510

2. Secondary Outcome: Mean Change From Baseline in Instantaneous Total Nasal Symptom Sscore (AM) for the Entire 14-day Study Period Compared to Placebo
Description: End of 24 hour dosing interval: This endpoint is change from baseline in instantaneous (tNSS) for the 14-day study period compared to placebo to observe if the duration of efficacy lasts 24 hours on a day to day basis. Instantaneous tNSS consists of runny nose, itchy nose, nasal congestion, and sneezing. Each symptom is rated on a scale from 0-3: 0=none, 1=mild, 2=moderate, and 3=severe.
  Least square means was controlled for study day as the within-patient effect, treatment group and site as the between-patient effects, treatment by-study day interaction, and baseline as a covariate.
Time Frame: baseline to 14 Days
Measure: Least Squares Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Astepro 0.15%
Number analyzed (Participants) | 255 | 251
Score on a scale | -0.83 (1.842) | -1.43 (2.088)
Statistical Analysis 1: Comparison: Placebo vs Astepro 0.15%; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA is being used due to a covariate being included in the model. The covariate is baseline TNSS score; Mean Difference (Final Values) = -0.6063, 95% CI [-0.94 to -0.27], Standard Error of Mean 0.1697

3. Secondary Outcome: Change From Baseline in Instantaneous Total Nasal Symptom Score for the Entire 14-day Study Period Compared to Placebo (AM and PM Combined)
Description: instantaneous (subjects rate how they feel "right now") total nasal symptom score consisting of runny nose, itchy nose, nasal congestion, and sneezing was assessed twice daily. Each symptom is rated on a scale from 0-3: 0=none, 1=mild, 2=moderate, and 3=severe. Total possible score is 24 per day.
  Least square means was controlled for study day as the within-patient effect, treatment group and site as the between-patient effects, treatment by-study day interaction, and basline as a covariate.
Time Frame: baseline to 14 Days
Measure: Least Squares Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Astepro 0.15%
Number analyzed (Participants) | 255 | 251
scores on a scale
  Baseline symptom score | 17.63 (3.906) | 17.43 (3.665)
  Overall change from baseline | -1.73 (3.669) | -3.12 (4.099)
Statistical Analysis 1: Comparison: Placebo vs Astepro 0.15%; Overall change from baseline; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA is being used due to a covariate being included in the model. The covariate is baseline TNSS score; Mean Difference (Final Values) = -1.3947, 95% CI [-2.06 to -0.73], Standard Error of Mean 0.3391

4. Secondary Outcome: Change From Baseline in 12-hour Reflective Total Ocular Symptom Score and Instantaneous Total Ocular Symptom Score for the Entire 14-day Study Period Compared to Placebo (AM and PM Combined)
Description: reflective and instantaneous symptom scores (itchy eyes, watery eyes and red eyes) were assessed twice daily. Each symptom is rated on a scale from 0-3: 0=none, 1=mild, 2=moderate, and 3=severe. Total possible TOSS score is 9 per day.
  Least square means was controlled for study day as the within-patient effect, treatment group and site as the between-patient effects, treatment by-study day interaction, and basline as a covariate.
Time Frame: baseline to14 Days
Measure: Least Squares Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Astepro 0.15%
Number analyzed (Participants) | 255 | 251
Scores on a scale
  Baseline: Reflective | 11.85 (4.580) | 11.52 (4.273)
  Change from Baseline: Reflective | -1.28 (2.932) | -2.21 (3.419)
  Baseline: Instantaneous | 11.33 (4.700) | 11.08 (4.449)
  Change from Baseline: Instantaneous | -1.05 (2.913) | -2.03 (3.313)
Statistical Analysis 1: Comparison: Placebo vs Astepro 0.15%; reflective TOSS change in baseline; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA is being used due to a covariate being included in the model. The covariate is baseline TNSS score; Mean Difference (Final Values) = -0.9284, 95% CI [-1.47 to -0.39], Standard Error of Mean 0.2741

5. Secondary Outcome: Change From Baseline to Visit 4 in the Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) Compared to Placebo in Subjects 18 Years of Age and Older
Description: A 28-item RQLQ was completed on Day 1 and Day 14 or Early temination. The RQLQ consists of 7 domains rated on a 7 point scale with 0 being not troubled by the allergy symptoms, and 6 being extremely troubled/all of the time.
  Scores for a series of subsclaes are not combined for a total overall score, rather domain score will be calculated from the mean score of all items in the domain. Overall score will be calculated from the mean score of all items.
Time Frame: 14 Days
Measure: Least Squares Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Placebo | Astepro 0.15%
Number analyzed (Participants) | 255 | 251
Units on a Scale
  Baseline: | 4.39 (1.149) | 4.33 (1.226)
  Change from Baseline: | -0.98 (1.463) | -1.33 (1.599)
Statistical Analysis 1: Comparison: Placebo vs Astepro 0.15%; change from baseline; Test type: Superiority or Other; p = 0.010, ANCOVA; ANCOVA is being used due to a covariate being included in the model. The covariate is baseline TNSS score

6. Secondary Outcome: Change From Baseline on Direct Visual Nasal Exams to 14 Days
Description: Examination of head and neck (scale: None, Mild, Moderate, Severe) for Epistaxis, Mucosal Edema, Nasal Discharge, Mucosal erythema, Mucosal Bleeding, and Crusting of mucosa. Nasal irratation was rated: 0 = None, Grade 1A = focal irritation, Grade 1B = superficial mucosal erosion, Grade 2 = moderate mucosal erosion,Grade 3 = ulceration, Grade 4 = septal perforation
Time Frame: baseline and 14 days
Measure: Number; unit: Participants
Arm/Group | Placebo | Astepro 0.15%
Number analyzed (Participants) | 255 | 251
Participants
  Epistaxis: screening - None (n=255, 251) | 255 | 249
  Epistaxis: screening - Mild (n=255, 251) | 0 | 2
  Epistaxis: screening - Moderate (n=255, 251) | 0 | 0
  Epistaxis: screening - Severe (n=255, 251) | 0 | 0
  Epistaxis: Day 14/ET - None (n=255, 249) | 254 | 246
  Epistaxis: Day 14/ET - Mild (n=255, 249) | 1 | 3
  Epistaxis: Day 14/ET - Moderate (n=255, 249) | 0 | 0
  Epistaxis: Day 14/ET - Severe (n=255, 249) | 0 | 0
  Nasal Irritation: screening - None (n=255, 251) | 236 | 231
  Nasal Irritation: screening -Grade 1A (n=255, 251 | 19 | 20
  Nasal Irritation: screening -Grade 1B (n=255, 251) | 0 | 0
  Nasal Irritation: screening - Grade 2 (n=255, 251) | 0 | 0
  Nasal Irritation: screening - Grade 3 (n=255, 251) | 0 | 0
  Nasal Irritation: screening - Grade 4 (n=255, 251) | 0 | 0
  Nasal Irritation: Day 14/ET - None(n=255, 249) | 246 | 228
  Nasal Irritation: Day 14/ET- Grade 1A (n=255, 249) | 8 | 19
  Nasal Irritation: Day 14/ET- Grade 1B (n=255, 249) | 1 | 2
  Nasal Irritation: Day 14/ET- Grade 2 (n=255, 249) | 0 | 0
  Nasal Irritation: Day 14/ET- Grade 3 (n=255, 249) | 0 | 0
  Nasal Irritation: Day 14/ET- Grade 4 (n=255, 249) | 0 | 0
  Mucosal Edema: screening - None (n=255, 251) | 18 | 19
  Mucosal Edema: screening - Mild (n=255, 251) | 54 | 58
  Mucosal Edema: screening - Moderate (n=255, 251) | 155 | 129
  Mucosal Edema: screening - Severe (n=255, 251) | 28 | 45
  Mucosal Edema: Day 14/ET - None (n=255, 249) | 18 | 24
  Mucosal Edema: Day 14/ET - Mild (n=255, 249) | 73 | 66
  Mucosal Edema: Day 14/ET - Moderate (n=255, 249) | 131 | 123
  Mucosal Edema: Day 14/ET - Severe (n=255, 249) | 33 | 36
  Nasal Discharge: screening - None (n=255, 251) | 41 | 33
  Nasal Discharge: screening - Mild (n=255, 251) | 102 | 108
  Nasal Discharge: screening - Moderate (n=255, 251) | 97 | 89
  Nasal Discharge: screening - Severe (n=255, 251) | 15 | 21
  Nasal Discharge: Day 14/ET - None (n=255, 249) | 38 | 45
  Nasal Discharge: Day 14/ET- Mild (n=255, 249) | 130 | 120
  Nasal Discharge: Day 14/ET - Moderate (n=255, 249) | 80 | 67
  Nasal Discharge: Day 14/ET - Severe (n=255, 249) | 7 | 17
  Mucosal Erythema: screening - None (n=255, 251) | 153 | 139
  Mucosal Erythema: screening -Mild (n=255, 251) | 49 | 60
  Mucosal Erythema: screening -Moderate (n=255, 251) | 47 | 49
  Mucosal Erythema: screening -Severe (n=255, 251) | 6 | 3
  Mucosal Erythema: Day 14/ET - None (n=255, 249) | 153 | 145
  Mucosal Erythema: Day 14/ET - Mild (n=255, 249) | 49 | 50
  Mucosal Erythema: Day 14/ET Moderate (n=255, 249) | 43 | 36
  Mucosal Erythema: Day 14/ET Severe (n=255, 249) | 10 | 18
  Mucosal Bleeding: screening - None (n=255, 251) | 251 | 247
  Mucosal Bleeding: screening - Mild (n=255, 251) | 4 | 3
  Mucosal Bleeding: screening Moderate (n=255, 251) | 0 | 1
  Mucosal Bleeding: screening - Severe (n=255, 251) | 0 | 0
  Mucosal Bleeding: Day 14/ET - None (n=255, 249) | 254 | 243
  Mucosal Bleeding: Day 14/ET - Mild (n=255, 249) | 1 | 6
  Mucosal Bleeding: Day 14/ET Moderate (n=255, 249) | 0 | 0
  Mucosal Bleeding: Day 14/ET - Severe (n=255, 249) | 0 | 0
  Crusting of Mucosa: screening - None (n=255, 251) | 236 | 229
  Crusting of Mucosa: screening - Mild (n=255, 251) | 17 | 19
  Crusting of Mucosascreening Moderate (n=255,251) | 2 | 3
  Crusting of Mucosa: screening Severe (n=255, 251) | 0 | 0
  Crusting of Mucosa: Day 14/ET - None (n=255, 249) | 248 | 240
  Crusting of Mucosa: Day 14/ET - Mild (n=255, 249) | 5 | 8
  Crusting of Mucosa:Day 14/ET Moderate (n=255, 249) | 1 | 1
  Crusting of Mucosa:Day 14/ET Severe (n=255, 249) | 1 | 0

ADVERSE EVENTS:
Arm/Group | Placebo | Astepro 0.15%
Serious Adverse Events (participants affected / at risk) | 0/255 | 0/251
Other Adverse Events (participants affected / at risk) | 2/255 | 25/251
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=255) | Astepro 0.15% (N=251)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 9 (9)
Dysgeusia (Nervous system disorders) | 2 (2) | 6 (6)
Headache (Nervous system disorders) | 0 (0) | 5 (5)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For multicenter studies, joint publication is required to assure that the initial publication is based on all data from all sites and investigators participating in these studies agree not to present data gathered individually or by subgroup centers before the initial publication unless jointly agreed by all other investigators and the sponsor. authorship will be determined by mutual agreement.